CLINICAL TRIAL: NCT01536093
Title: Oropharyngeal Administration of Colostrum to Extremely Low Gestational Age Newborns
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OAC-01-ELGAN
Record Dates: First submitted 2012-01-06; First posted 2012-02-20 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Extremely Low Gestational Age Newborn; Premature Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colostrum (Experimental): oropharyngeal administration of own mother's colostrum
  Interventions: Other: oropharyngeal administration of own mother's colostrum
- Placebo (Placebo Comparator): oropharyngeal administration of sterile water
  Interventions: Other: oropharyngeal administration of sterile water

INTERVENTIONS:
Other: oropharyngeal administration of own mother's colostrum — application of 0.2 mL of colostrum to the infant's oropharyngeal mucosa every 3 hours for 3 days from the postnatal 48 to 96 hours.
  Arms: Colostrum
Other: oropharyngeal administration of sterile water — application of 0.2 mL of sterile water to the infant's oropharyngeal mucosa every 3 hours for 3 days from the postnatal 48 to 96 hours.
  Arms: Placebo

SUMMARY:
Colostrum is rich in cytokines and other immune agents that may provide immunomodulatory protection against nosocomial infection in extremely premature infants. However, most of them could not proceed enteral feedings due to clinical instability in the first few days. Recent studies supports oropharyngeal administration as a potentially safe and effective delivery method for immunologic benefits and only small amount of colostrum could be administrated for immune therapy for extremely premature babies. The purpose of this study is to determine the beneficial effects of oropharyngeal administration of colostrum for immunologic aspects in extremely low gestational age infants and evaluated the safety of this method to extremely premature infants in the first few days of life.

ELIGIBILITY:
Inclusion Criteria:

* premature infant with a gestational age less than 28 weeks born at Seoul National University Hospital and admit to the Seoul National University Children's Hospital NICU immediately after birth
* parents of the infant signed to the informed consent form with voluntary agreement

Exclusion Criteria:

* infants with major congenital anomalies or chromosomal syndromes
* infants of mothers not willing to provide colostrum in the first week of life
* infants of mothers with known infectious diseases that may be transmitted through the breast milk such as HIV, hepatitis C or active TB

Ages: 48 Hours to 96 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee J, Kim HS, Jung YH, Choi KY, Shin SH, Kim EK, Choi JH. Oropharyngeal colostrum administration in extremely premature infants: an RCT. Pediatrics. 2015 Feb;135(2):e357-66. doi: 10.1542/peds.2014-2004. PMID 25624376

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colostrum | Placebo
Started | 24 | 24
Completed | 21 | 21
Not Completed | 3 | 3
Not completed — Death | 1 | 2
Not completed — absence of maternal colostrum | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colostrum | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational Age
  weeks | 26.1 (1.4) | 26.0 (1.4) | 26.1 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 11 | 10 | 21
Birth weight [Mean (Standard Deviation); unit: g] | 862.2 (234.8) | 842.4 (250.4) | 849.3 (239.8)

OUTCOME MEASURES:

1. Primary Outcome: Urinary Secretary IgA Concentration at 2 Weeks of Age
Time Frame: 2 weeks of age
Measure: Mean (Standard Deviation); unit: ng per g creatinine
Arm/Group | Colostrum | Placebo
Number analyzed (Participants) | 21 | 21
ng per g creatinine | 233.8 (37.4) | 48.3 (24.1)
Statistical Analysis 1: Comparison: Colostrum vs Placebo; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Urinary Secretary IgA Concentration at 1 Week of Age
Time Frame: 1 week of age
Measure: Mean (Standard Deviation); unit: ng per g creatinine
Arm/Group | Colostrum | Placebo
Number analyzed (Participants) | 21 | 21
ng per g creatinine | 71.4 (33.1) | 26.5 (6.7)
Statistical Analysis 1: Comparison: Colostrum vs Placebo; Test type: Superiority or Other; p = 0.043, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Salivary TGF-beta 1 Concentration at 2 Week of Age
Time Frame: 2 week of age
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Colostrum | Placebo
Number analyzed (Participants) | 21 | 21
ug/mL | 39.2 (6.3) | 69.7 (12.7)
Statistical Analysis 1: Comparison: Colostrum vs Placebo; Test type: Superiority or Other; p = 0.032, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Salivary IL-8 Concentration at 2 Weeks of Age
Time Frame: 2 weeks of age
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Colostrum | Placebo
Number analyzed (Participants) | 21 | 21
ng/mL | 2.58 (1.01) | 4.90 (1.19)
Statistical Analysis 1: Comparison: Colostrum vs Placebo; Test type: Superiority or Other; p = 0.038, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Concentration of Urinary Lactoferrin
Time Frame: 1 week of age
Measure: Mean (Standard Deviation); unit: ug per g creatinine
Arm/Group | Colostrum | Placebo
Number analyzed (Participants) | 21 | 21
ug per g creatinine | 3.51 (1.32) | 0.98 (0.28)
Statistical Analysis 1: Comparison: Colostrum vs Placebo; Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Concentration of Urinary IL-1 Beta
Time Frame: 2 weeks of age
Measure: Mean (Standard Deviation); unit: ug per g creatinine
Arm/Group | Colostrum | Placebo
Number analyzed (Participants) | 21 | 21
ug per g creatinine | 55.25 (7.12) | 91.80 (11.86)
Statistical Analysis 1: Comparison: Colostrum vs Placebo; Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Concentration of Salivary Lactoferrin, Lysozyme, Alpha-lactalbumin and Cytokines
Time Frame: 1 week of age
Reporting Status: Not Posted

8. Secondary Outcome: Concentration of Salivary Lactoferrin, Lysozyme, Alpha-lactalbumin and Cytokines
Time Frame: 2 weeks of age
Reporting Status: Not Posted

9. Secondary Outcome: Time to Reach Full Feeding
Description: day of life when the baby reaches full enteral feeding, defined as a volume above 120~130mL/kg/day
Time Frame: up to 2 months of age
Reporting Status: Not Posted

10. Secondary Outcome: Total Hospital Admission Duration
Description: days from admission to discharge from NICU
Time Frame: up to 4 months of age
Reporting Status: Not Posted

11. Secondary Outcome: Episodes of Culture Positive Sepsis
Description: numbers of documented sepsis events defined as isolation of the microorganism from ≥ 1 blood culture + ≥ 1 clinical symptoms or sign (fever, hypothermia, apnea, bradycardia, hypo-/hyperglycemia)
Time Frame: from date of randomization up to 4 months of age
Reporting Status: Not Posted

12. Secondary Outcome: Episodes of Necrotizing Enterocolitis ≥ Bell's Stage 2
Time Frame: from date of randomization up to 4 months of age
Reporting Status: Not Posted

13. Secondary Outcome: Episodes of Pneumonia
Description: numbers of documented pneumonia events those accompanied with increased tracheal secretion, increased ventilatory setting and treated with antibiotics
Time Frame: from date of randomization up to 4 months of age
Reporting Status: Not Posted

14. Secondary Outcome: Development of Bronchopulmonary Dysplasia ≥ Moderate
Time Frame: up to 4 months of age
Reporting Status: Not Posted

15. Secondary Outcome: Development of Intraventricular Hemorrhage ≥ Grade 3
Time Frame: up to 4 months of age
Reporting Status: Not Posted

16. Secondary Outcome: In-hospital Death
Time Frame: up to 4 months of age
Reporting Status: Not Posted

17. Secondary Outcome: Development of Adverse Effects
Description: category of adverse effects
  1. general - fever or hypothermia, rash
  2. respiratory & cardiovascular - apnea, tachypnea, desaturation, hypotension, bradycardia, tachycardia
  3. gastrointestinal - abdominal distension, bilious gastric remain, vomiting, bloody stool, necrotizing enterocolitis
  4. renal - oliguria (urine output < 1.0cc/kg/day)
  5. laboratory - hypo-/hyper-natremia, acidosis, hypercarbia
Time Frame: from the start date of oropharyngeal administration of colostrum or sterile water to 1 week of age
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Colostrum | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No